CLINICAL TRIAL: NCT03428477
Title: A Randomised Placebo-controlled Phase III Trial of the Effect of the Omega-3 Fatty Acid Eicosapentaenoic Acid (EPA) on Colorectal Cancer Recurrence and Survival After Surgery for Resectable Liver Metastases
Brief Title: EPA for Metastasis Trial 2
Acronym: EMT2
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Mark A Hull, PhD FRCP (Other)
Collaborators: Yorkshire Cancer Research (Other); Amarin Pharma Inc. (Industry)
Responsible Party: Sponsor-Investigator, Mark A Hull, PhD FRCP, Prof Mark Hull, University of Leeds
Organization: University of Leeds (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MO16/053
Record Dates: First submitted 2018-01-11; First posted 2018-02-09 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Liver Metastasis; Colon Cancer
Keywords: Liver metastases; Colon Cancer
MeSH Terms: conditions — Colonic Neoplasms | interventions — eicosapentaenoic acid ethyl ester

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Icosapent Ethyl (EPA-EE) (Experimental): Soft gelatin capsules containing 1g pure EPA-EE equivalent to 914mg EPA-FFA. Administered as 4g per day to be taken as 2 capsules in the morning and 2 capsules in the evening.
  Interventions: Drug: Icosapent Ethyl
- Placebo (Placebo Comparator): Soft gelatin capsules containing light mineral oil. 4 capsules to be taken per day (2 in the morning and 2 in the evening).
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Icosapent Ethyl — Composition: soft amber to light yellow, oblong gelatin capsules. One capsule contains 1g pure EPA-EE Dose: 4 capsules per day
  Other Names: Vascepa
  Arms: Icosapent Ethyl (EPA-EE)
Other: Placebo — Composition: soft, amber to light yellow, oblong gelatin capsules containing light mineral oil:
  Dose: 4 capsules per day
  Arms: Placebo

SUMMARY:
A significant proportion of patients who undergo liver surgery to remove bowel cancer that has spread to the liver (metastases) develop disease recurrence and die from the disease. A previous small study (the EMT study) suggested a possible survival benefit in patients who took the naturally-occurring omega-3 fatty acid EPA (a fish oil supplement) before liver surgery. The EMT2 study is a larger study which will recruit 448 men and women with liver metastases from bowel cancer. Trial participants will receive either Icosapent Ethyl (pure EPA derived from fish oil) or placebo (dummy capsules). EMT2 will investigate whether patients who take this supplement before liver surgery and for up to four years after surgery, remain free of recurrence for longer than those who take placebo (dummy capsules)

DETAILED DESCRIPTION:
Despite significant advances in diagnosis and treatment of colorectal cancer (CRC), it remains the second most common cause of cancer-related death in the UK. The majority of deaths from CRC are related to distant metastasis, predominantly to the liver. Overall 5-year survival following liver resection and adjuvant chemotherapy for colorectal cancer liver metastases (CRCLM) is, at best, 40-60%. Despite surgery with curative intent, up to 60% of patients develop recurrence within 2 years of surgery. The preliminary EMT study was a Phase II RCT of EPA 2 g daily in patients (n=88) undergoing liver resection surgery for CRCLM. Although there was no difference in the primary endpoint (tumour proliferation index), metastases from the EPA arm had a lower vascularity score (suggesting possible anti-angiogenic activity) than placebo-treated tumours. Although EPA (or placebo) treatment was limited to the pre-operative period, overall survival (OS) and disease-free survival (DFS) were specified as exploratory end-points on the basis that oral dosing with EPA before liver surgery would provide tissue EPA exposure in the immediate peri-operative period with prolonged bioavailability in the post-operative period due to the slow tissue 'washout' kinetics of EPA. Survival analysis demonstrated that the median DFS in the EPA group was 22.6 months compared with 14.7 months in the placebo group. Any DFS benefit was explained by a reduction in CRC recurrence from 12 months after surgery onwards.

The EMT2 study is a randomised, double-blind, placebo-controlled, multi-centre, phase III trial of the omega-3 fatty acid (O3FA) eicosapentaenoic acid (EPA) as the ethyl ester (icosapent ethyl [IPE; Vascepa®]) in patients undergoing liver resection surgery for colorectal cancer liver metastasis (CRCLM) with curative intent designed to determine whether EPA treatment improves Progression-Free Survival (PFS). A key secondary objective is overall survival (OS).

Investigators will recruit adult individuals listed for CRCLM resection with curative intent.

Randomisation will be 1:1 to receive either IPE capsules or placebo capsules. 4 capsules per day containing IPE (equivalent to 4 g EPA-ethyl ester [EE] daily) or 4 placebo capsules per day. Participants will start treatment a prior to CRCLM surgery and will continue to receive treatment for a minimum of 2 years and a maximum of 4 years post-liver resection. Participants are followed up for 60 days beyond the end of treatment.

Participants are clinically assessed 6 months post-operatively (from liver resection) and at 6-monthly intervals thereafter for disease progression/recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18 years
* Able to provide written informed consent
* Histological diagnosis of colorectal cancer with evidence of liver metastases
* Planned liver resection surgery for colorectal cancer liver metastases with curative intent, including repeat 're-do' colorectal cancer liver metastases surgery (a second independent resection for a separate colorectal cancer liver recurrence)
* Intention to receive IMP prior to colorectal cancer liver metastases surgery

Exclusion Criteria:

* Previous CRCLM surgery for the management of the current metastatic disease
* Incurable extra-hepatic metastases
* Current (in the last 2 months) or planned regular (>3 doses per week) use of O3FA-containing drugs or supplements, including Vazkepa®, Omacor®, fish oil and cod-liver oil supplements
* Fish/seafood allergy
* Diagnosis of hereditary fructose intolerance
* Soya or peanut allergy
* Inability to comply with trial treatment and follow-up schedule
* Known bleeding tendency/condition (e.g. von Willebrand disease)
* A previous malignancy within the last 5 years other than:

  * colorectal cancer
  * non-melanoma skin cancer where treatment consisted of resection only or radiotherapy
  * ductal carcinoma in situ (DCIS) where treatment consisted of resection only
  * cervical carcinoma in situ where treatment consisted of resection only
  * superficial bladder carcinoma where treatment consisted of resection only
* A previous malignancy where the patient has been disease free for ≤ 5 years
* Pregnant or breastfeeding women or women of childbearing potential not willing to use effective contraceptive measures. Women of childbearing potential are defined as fertile, following menarche and until becoming post-menopausal, unless permanently sterile
* Men defined as fertile (post-pubescent and not permanently sterile by vasectomy or bilateral orchidectomy) and not willing to use effective contraceptive measures if appropriate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 418 (Actual)
Dates: Start 2018-05-02 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | Minimum of 2 years follow-up
  PFS is defined as the time from randomisation to death (from any cause), first documented evidence of disease progression, new recurrence or clinical deterioration unequivocally due to disease progression

SECONDARY OUTCOMES:
Overall Survival (OS) | Minimum of 2 years follow-up
  The time from randomisation to death, from any cause (key secondary endpoint)
Safety and Tolerability of Icosapent Ethyl | Minimum of 2 years follow-up
  The number of participants with treatment-emergent adverse events as defined by CTCAE v4.0
Patient reported quality of life 1 | Minimum of 2 years follow-up
  Measured using the EQ-5D questionnaire
Patient reported quality of life 2 | Minimum of 2 years follow-up
  Measured using the EORTC QLQ-C30 questionnaire
Patient reported quality of life 3 | Minimum of 2 years follow-up
  Measured using the QLQ-LMC21 questionnaire
New Primary Cancers | Minimum of 2 years follow-up
  Excluding DCIS, cervical carcinoma in situ, superficial bladder carcinoma where treatment consisted of resection only and non-melanoma skin cancer where treatment consisted of resection or radiotherapy only)

OTHER OUTCOMES:
Red Blood Cell Membrane EPA content (exploratory endpoint) | Samples taken at baseline, surgery and 6 months after surgery
  EPA content measured at baseline, surgery and 6 months after surgery. Samples taken at selected sites only
Change in lean body mass (exploratory endpoint) | 6 months and up to 4 years follow up
  Change in lean body mass measured by CT scanning during follow-up as assessed by the L3 skeletal muscle index score. Scans reviewed from selected sites only

CONTACTS AND LOCATIONS:
Overall Officials: Mark Hull, Principal Investigator — University of Leeds
Locations (13):
- United Kingdom (13):
  - Oxford University Hospital NHS Foundation Trust, Oxford, Oxfordshire
  - Hampshire Hospitals NHS Foundation Trust, Basingstoke, Royal Hampshire
  - Aintree University Hospitals NHS Foundation Trust, Aintree
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham
  - Cambridge UniversityHospitals NHS Foundation Trust, Cambridge
  - University Hospital of Wales, Cardiff
  - Leeds Teaching Hospitals NHS Foundation Trust, Leeds
  - King's College London, London
  - Royal Free London NHS Foundation Trust, London
  - Newcastle Upon Tyne Hospitals NHS Foundation Trust, Newcastle
  - Nottingham University Hospitals NHS Trust, Nottingham
  - Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield
  - University Hospital Southampton NHS Foundation Trust, Southampton

IPD SHARING:
Plan to Share IPD: Yes
The datasets generated during the current study will be available upon request from the Clinical Trials Research Unit at the University of Leeds.
  De-identified individual participant data datasets generated during the current study will be available upon request from the Clinical Trials Research Unit, University of Leeds (contact CTRU-DataAccess@leeds.ac.uk in the first instance).
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be made available at the end of the trial, i.e. usually when all primary and secondary endpoints have been met and all key analyses are complete. Data will remain available from then on, for as long as CTRU retains the data.
Access Criteria: Data will be released for secondary research purposes, where the Chief Investigator, Sponsor and CTRU agree that the proposed use has scientific value and will be carried out to a high standard (scientific rigour and information governance and security), and that suitable resources are available. Data will be released in line with participants' consent, all applicable laws relating to data protection and confidentiality, and any contractual obligations to which the CTRU is subject. No IPD will be released before an appropriate agreement is in place governing data retention, usually stipulating that data recipients must delete their copy of the data at the end of the project.
  The CTRU believes it is best practice for researchers who generated datasets to be involved in subsequent uses of those datasets. Recipients of trial data for secondary research will also receive data dictionaries, key trial documents and any other information required to reuse the datasets.

REFERENCES:
- [Derived] Hull MA, Ow PL, Ruddock S, Brend T, Smith AF, Marshall H, Song M, Chan AT, Garrett WS, Yilmaz O, Drew DA, Collinson F, Cockbain AJ, Jones R, Loadman PM, Hall PS, Moriarty C, Cairns DA, Toogood GJ. Randomised, placebo-controlled, phase 3 trial of the effect of the omega-3 polyunsaturated fatty acid eicosapentaenoic acid (EPA) on colorectal cancer recurrence and survival after surgery for resectable liver metastases: EPA for Metastasis Trial 2 (EMT2) study protocol. BMJ Open. 2023 Nov 29;13(11):e077427. doi: 10.1136/bmjopen-2023-077427. PMID 38030258

DOCUMENTS (1):
  • Study Protocol (2022-07-27): https://cdn.clinicaltrials.gov/large-docs/77/NCT03428477/Prot_003.pdf